CLINICAL TRIAL: NCT05729789
Title: Investigating Group Written Exposure Therapy for Posttraumatic Stress Disorder: A Pilot Study
Brief Title: Group Written Exposure Therapy for Posttraumatic Stress Disorder
Acronym: GWET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Jenna Boyd, Dr. Jenna Boyd, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15477
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: cognitive behavioural therapy; written exposure therapy; group therapy; posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group Written Exposure Therapy (Experimental): Patients will be invited to participate in group Written Exposure Therapy (described in the "Interventions" section).
  Interventions: Behavioral: Group Written Exposure Therapy

INTERVENTIONS:
Behavioral: Group Written Exposure Therapy — Group Written Exposure Therapy (GWET) is a brief cognitive behavioural therapy for PTSD aimed at allowing patients to process their traumatic experiences in a safe environment. GWET will consist of 6 group sessions (1 orientation session and 5 weekly group sessions). Participants will be asked to complete weekly in-session written exposures where they will recount their traumatic experience. The written exposure will be followed by a guided discussion about the experience of writing the exposure. There is no homework assigned between sessions. However, group members will be asked to refrain from avoiding thinking about the trauma between sessions.

SUMMARY:
The goal of this clinical trial is to test if Written Exposure Therapy (WET) works well in a group setting in patients with post-traumatic stress disorder (PTSD).

The main questions it aims to answer are:

* Does group WET lead to a reduction in symptoms of PTSD?
* Is group WET better at reducing the number of patients that drop out of treatment in comparison to group Cognitive Processing Therapy (CPT)?

Participants will:

* Attend 6 weekly sessions of group WET that will be delivered online by two therapists (psychologist and social worker)
* Complete questionnaires relating to their symptoms at different points throughout the treatment

Researchers will evaluate change in PTSD symptoms over time for people who participate in group WET. They will also compare the results of group WET to the results of group CPT to see if group WET shows a similar reduction in symptoms of PTSD and fewer treatment drop-outs.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effectiveness of group WET (G-WET) in reducing symptoms of PTSD in an outpatient hospital setting. In order to do so, we will evaluate outcomes of G-WET from pre- to post-treatment and at one month follow-up. We will also compare outcomes of G-WET to published benchmarks of individual WET outcomes and to a representative cohort of individuals who participate in group CPT at our clinic. A secondary aim of the study is to evaluate attendance and drop-out rates for group WET. In order to achieve this, we will recruit a sample of 63 individuals between the ages of 18 and 65 to participate in a group WET 6-session protocol (1 orientation session and 5 WET sessions) from an outpatient anxiety and related disorders clinic waitlist for group CPT. Participants will complete measures assessing PTSD, related symptoms (e.g., depression, anxiety) and group cohesion at pre-treatment, post-treatment, and 1-month follow-up. Attendance and drop-out rates will also be recorded. We hypothesize that group WET will be associated with significant reductions in PTSD symptoms and related symptoms and low dropout rates (i.e., less than 10%). We also hypothesize that outcomes for group WET will be comparable to those for group CPT and published individual WET benchmarks.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and older
* Diagnosis of PTSD
* Able to provide written informed consent and can read and write in English

Exclusion Criteria:

* Diagnosis of an active severe substance use disorder (SUD)
* Diagnosis of a psychotic disorder (schizophrenia, schizoaffective disorder, etc.)
* Untreated active psychotic, manic or hypomanic symptoms
* Has attempted suicide in the 2 months prior to beginning treatment
* Has engaged in high-risk self-harm (e.g., cutting, burning, asphyxiation) in the 2 months prior to beginning treatment
* Has completed CPT in the past
* Has completed another active PTSD treatment, such as Prolonged Exposure or EMDR within the last year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-05-09 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the PTSD Checklist for DSM-5 (PCL-5) | Weekly at each group session, 1 week before treatment begins, 1 week after treatment ends, and 1-month follow-up.
  20-item self-report questionnaire assessing symptoms of PTSD over the past week.

SECONDARY OUTCOMES:
Change from baseline on the Posttraumatic Cognitions Inventory (PTCI) | 1 week before treatment begins, 1 week after treatment ends, and 1-month follow-up.
  36-item self-report questionnaire assessing negative beliefs across three subscales: negative cognitions about the self, negative cognitions about the world, and self-blame.
Change from baseline on the Depression, Anxiety, Stress Scale -21 Item Version (DASS-21) | 1 week before treatment begins, 1 week after treatment ends, and 1-month follow-up.
  21-item self-report measure with three subscales measuring depression, anxiety, and stress symptoms.
Change from baseline on the Difficulties in Emotion Regulation Scale (DERS) | 1 week before treatment begins, 1 week after treatment ends, and 1-month follow-up.
  36-item self-report measure assessing emotion regulation difficulties.
Change from baseline on the Illness Intrusiveness Rating Scale (IIRS) | 1 week before treatment begins, 1 week after treatment ends, and 1-month follow-up.
  13-item self-report measure assessing the effect of illness on domains of quality of life.
Group Cohesion Scale-Revised (GCS-R) | 1 week after treatment ends.
  Self-report measure assessing group member's perception of their group and the strength of the bonds formed.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Boyd, Ph.D., Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- Anxiety Treatment and Research Clinic, St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sloan DM, Marx BP, Resick PA, Young-McCaughan S, Dondanville KA, Straud CL, Mintz J, Litz BT, Peterson AL; STRONG STAR Consortium. Effect of Written Exposure Therapy vs Cognitive Processing Therapy on Increasing Treatment Efficiency Among Military Service Members With Posttraumatic Stress Disorder: A Randomized Noninferiority Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2140911. doi: 10.1001/jamanetworkopen.2021.40911. PMID 35015065
- [Background] Sloan, D.M., & Marx, B.P. (2019). Written exposure therapy for PTSD: A brief treatment approach for mental health professionals. American Psychological Association.
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Background] Antony, M.M., Bieling, P.J., Cox, B.J., Enns, M.W., & Swinson, R.P. (1998). Psychometric properties of the 42-item and 21-item versions of the Depression Anxiety Stress Scales in clinical groups and a community sample. Psychological Assessment, 10(2), 176-181.
- [Background] Foa, E.B., Ehlers, A., Clark, D.M., Tolin, D.F., & Orsillo, S.M. (1999). The Posttraumatic Cognitions Inventory (PTCI): Development and validation. Psychological Assessment, 11(3), 303-314.
- [Background] Devins GM. Using the illness intrusiveness ratings scale to understand health-related quality of life in chronic disease. J Psychosom Res. 2010 Jun;68(6):591-602. doi: 10.1016/j.jpsychores.2009.05.006. Epub 2009 Jul 17. PMID 20488277
- [Background] Treadwell, T., Lavertue, N., Kumar, V. K., & Veeraraghavan, V. (2001). The Group Cohesion Scale-Revised: Reliability and validity. International Journal of Action Methods: Psychodrama, Skill Training, and Role Playing, 54(1), 3-12.